CLINICAL TRIAL: NCT01493466
Title: Serum Proteomics Analysis for Dynamic Changes of Differential Proteins in Sepsis Patient With iTRAQ Labeling and LC-MS/MS
Brief Title: Serum Proteomics Analysis for Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Other Study IDs: 20111013-007(2); 2009BAI86B03 (Other Grant/Funding Number: Chinese National Science & Technology Pillar Program)
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: SIRS; Sepsis; Severe Sepsis; Death
Keywords: proteomics,; serum,; sepsis,; potential biomarkers,; dynamic changes; normal
MeSH Terms: conditions — Sepsis; Death

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Normal: normal person under physical examination
- SIRS: 1. temperature >38 ℃ or <36℃;
  2. pulse rate>90 beats/min;
  3. ventilatory rate>20 breaths/min or hyperventilation with partial pressure of arterial carbon dioxide (PaCO2)<32mmHg;
  4. white blood cell count>12,000μL-1 or <4000μL-1 or >10% immature cells
- spesis: sepsis is defined as SIRS plus confirmed infection.
- severe sepsis: 1. severe sepsis: sepsis associated with organ dysfunction, hypoperfusion, or hypotension;
  2. septic shock: sepsis with arterial hypotension, despite adequate ﬂuid resuscitation.
- death: sepsis patients within 48 hours before death

SUMMARY:
Serum proteomics is a very useful tool to identify various disease. The purpose of the present study was to find differential proteins among patient with normal, SIRS, sepsis, severe sepsis, death and to screen potential biomarkers for their dynamic changes. Serum proteins were identified by iTRAQ labeling and LC-MS/MS. The bioinformatics analysis was performed with the Mascot software and the International Protein Index (IPI) and the Gene Ontology (GO) Database and KEGG pathway Database. The differentially expressed proteins were verified by Western blot by another sample collected from clinical.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 years old and over;
* clinically confirmed infection;
* fulfilled at least two criteria of systemic inflammatory response syndrome
* (a) core temperature higher than 38 °C or lower than 36 °C
* (b)respiratory rate above 20/min, or PCO2 below 32 mmHg
* (c) pulse rate above 90/min, and
* (d) white blood cell count greater than 12,000/μl or lower than < 4,000/μl or less than 10% of bands.

Exclusion Criteria:

* younger than 18 years of age;
* acquired immunodeficiency syndrome;
* reduced polymorphonuclear granulocyte counts (< 500 μL-1);
* died within 24h after admission into the ICU, or refused to participate in the study, or declined treatment during the period of observation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects were selected from among inpatients who were hospitalized between May 2010 and Mar 2012 in the Respiratory ICU, Surgical ICU, and Emergency ICU, Chinese People's Liberation Army (CPLA) General Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Survival status | 28 days after admission to ICU
  The survival time of patients more than 28days is defined as survival. The survival time of patients less than 28days is defined as death.

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, MD, Study Director — Department of Respiratory Diseases, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijin, Beijing Municipality, China

REFERENCES:
- [Derived] Su L, Pan P, Yan P, Long Y, Zhou X, Wang X, Zhou R, Wen B, Xie L, Liu D. Role of vimentin in modulating immune cell apoptosis and inflammatory responses in sepsis. Sci Rep. 2019 Apr 5;9(1):5747. doi: 10.1038/s41598-019-42287-7. PMID 30952998